CLINICAL TRIAL: NCT01010893
Title: Tolerability and Immunogenicity Study of FLUVAL P Monovalent Influenza Vaccine in Adults and Elderly Persons
Brief Title: Tolerability and Immunogenicity of Fluval P Monovalent Influenza Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fluart Innovative Vaccine Ltd, Hungary (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FLUVAL P-H-06
Record Dates: First submitted 2009-11-07; First posted 2009-11-10 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Influenza
Keywords: pandemic; prevention; influenza; infection; influenza vaccine; vaccine; influenza in humans
MeSH Terms: conditions — Influenza, Human; Infections | interventions — Vaccination; Influenza Vaccines; Pandemics; Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Influenza vaccination (Experimental): Vaccination with Fluval P monovalent influenza vaccine with 6 μg HA/0.5 ml active ingredient content and aluminium phosphate gel adjuvant (dose: 0.5 ml /total 6 μg HA/ in both age groups, single dose).
  Interventions: Biological: Vaccination with Fluval P monovalent influenza vaccine
- Influenza vaccination and co-vaccination (Experimental): Vaccination with Fluval P monovalent influenza vaccine with 6 μg HA/0.5 ml active ingredient content and aluminium phosphate gel adjuvant (dose: 0.5 ml /total 6 μg HA/ in both age groups, single dose) AND with Fluval AB trivalent influenza vaccine with 15 μg HA/0.5ml/strain active ingredient content and aluminium phosphate gel adjuvant (dose: 0.5 ml /total 3x15 μg HA/ in both age groups, single dose).
  Interventions: Biological: Vaccination with Fluval P and Fluval AB influenza vaccines

INTERVENTIONS:
Biological: Vaccination with Fluval P and Fluval AB influenza vaccines — Vaccination with Fluval P monovalent influenza vaccine with 6 μg HA/0.5 ml active ingredient content and aluminium phosphate gel adjuvant (dose: 0.5 ml /total 6 μg HA/ in both age groups, single dose) AND with Fluval AB trivalent influenza vaccine with 15 μg HA/0.5ml/strain active ingredient content and aluminium phosphate gel adjuvant (dose: 0.5 ml /total 3x15 μg HA/ in both age groups, single dose).
  Other Names: Influenza; Pandemic vaccine; Seasonal vaccine; Co-vaccination; Prevention; Innfluenza vaccine; Influenza in humans
  Arms: Influenza vaccination and co-vaccination
Biological: Vaccination with Fluval P monovalent influenza vaccine — Fluval P monovalent influenza vaccine with 6 μg HA/0.5 ml active ingredient content and aluminium phosphate gel adjuvant
  Other Names: pandemic; influenza; prevention; vaccine; influenza vaccine; influenza in humans
  Arms: Influenza vaccination

SUMMARY:
To determine the tolerability and immunogenicity of FLUVAL P monovalent influenza vaccine in adults and elderly people, with the objective to verify efficacy and tolerability of the study drug.

DETAILED DESCRIPTION:
Primary Objective:

To assess tolerability/safety (incidence of adverse events) of the study drug. To assess the efficacy (immunogenicity) of the study drug by serology testing of blood samples taken at Day 21-28 after immunization in groups and age groups.

Secondary Objectives:

To assess the long-term safety of the study drug 50-60 days after immunization. To determine the tolerability of simultaneous administration of FLUVAL P monovalent pandemic influenza vaccine and FLUVAL AB trivalent seasonal influenza vaccine in case of adults and elderly people.

To assess the efficacy of the study drug by optional epidemiological follow-up of the participants until the end of the influenza season.

To assess the immunogenicity of the study drug by optional cross-reactive immunity tests performed with non-homologous influenza A and B virus strains.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 60 years, elderly people aged over 60 years, from both sexes, with full contractual capacity;
* Are in good health (as determined by vital signs and existing medical condition) or are in stable medical condition. Subjects will not be excluded with known adequately treated clinically significant organ or systemic diseases (e.g. asthma or diabetes), such that, in the opinion of the investigator, the significance of the disease will not compromise the subject's participation in the study;
* Femal volunteers of childbearing potential with a negative result from the urine pregnancy test prior to vaccination who agrees to use an acceptable contraception method or abstinence throughout the trial and not become pregnant for the duration of the study.
* Capable of understanding and complying with study protocol requirements;
* The volunteers provide written informed consent prior to initiation of study procedures;
* Absence of existence of any exclusion criteria.

Exclusion Criteria:

* Pregnancy or breast feeding or positive urine pregnancy test at baseline prior to vaccination;
* Known allergy to eggs or other components of the vaccine (in particular mercury);
* History of Guillain-Barré syndrome;
* Active neoplasm;
* Immunosuppressive therapy in the preceding 36 months;
* Concomitant corticosteroid therapy, including high-dose inhaled corticosteroids;
* Immunoglobulin (or similar blood product) therapy within 3 months prior to vaccination;
* Documented HIV, HBV or HCV infection;
* Chronic illness that, in the opinion of the investigator, may interfere with the evaluation of the immunoresponse;
* Acute febrile respiratory illness within one week prior to vaccination;
* Vaccine therapy within 4 weeks prior to vaccination;
* Influenza vaccination within 6 months prior to vaccination;
* Experimental drug therapy within 1 month prior to vaccination;
* Past or current psychiatric disease of the volunteer that upon judgement of the investigator may have effect on the objective decision-making of the volunteer;
* Alcohol or drug abuse of the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2009-08; Primary Completion 2009-09 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Post vaccination HI antibody titer | 21-28 days after vaccination
Incidence of adverse reactions | 21-28 days after vaccination

SECONDARY OUTCOMES:
Incidence of adverse reactions | 50-60 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Ferenc Tamas, MD, Principal Investigator — Pilisvorosvar District Doctor's Office; Anna Osi, Dr., Study Director — Omninvest Ltd.
Locations (2):
- Hungary (2):
  - District Doctor's Office, Pilisvörösvár
  - Fourmed Kft. Gyogyhaz, Veszprém

REFERENCES:
- [Derived] Vajo Z, Tamas F, Sinka L, Jankovics I. Safety and immunogenicity of a 2009 pandemic influenza A H1N1 vaccine when administered alone or simultaneously with the seasonal influenza vaccine for the 2009-10 influenza season: a multicentre, randomised controlled trial. Lancet. 2010 Jan 2;375(9708):49-55. doi: 10.1016/S0140-6736(09)62039-0. Epub 2009 Dec 15. PMID 20018367